CLINICAL TRIAL: NCT05771766
Title: Effects of Postural Drainage With and Without Aerobic Training on Respiratory Rate, Oxygen Saturation and Endurance in Chronic Suppurative Lung Disease
Brief Title: Postural Drainage With and Without Aerobic Training on Chronic Suppurative Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR& AHS/22/0737
Record Dates: First submitted 2023-01-04; First posted 2023-03-16 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Lung Disease Chronic
Keywords: CSLD, Respiratory Rate, Endurance, Oxygen Saturation
MeSH Terms: interventions — Drainage, Postural

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postural Drainage with Aerobic Training (Experimental): The intervention group will undergo Postural Drainage and additional Aerobic Training thrice a week for two weeks as well along with postural drainage. Aerobic training will include a 5-step stair-climbing and 10-step walk during each session.
  Interventions: Other: Postural Drainge and aerobic training
- Postural Drainage (Active Comparator): the group will receive postural drainage as baseline treatment thrice a week for two weeks.
  Interventions: Other: Postural Drainage

INTERVENTIONS:
Other: Postural Drainge and aerobic training — This will be a randomized controlled trial Patients will be divided into two groups randomly. Both groups will receive postural drainage as baseline treatment thrice a week for two weeks. The intervention group will undergo additional Aerobic Training thrice a week for two weeks as well along with postural drainage. Aerobic training will include 5-step stair-climbing and 10 step walk during each session.
  Arms: Postural Drainage with Aerobic Training
Other: Postural Drainage — Postural Drainage
  Arms: Postural Drainage

SUMMARY:
This will be a randomized controlled trial Patients will be divided into two groups randomly. Both groups will receive postural drainage as baseline treatment thrice a week for two weeks. The intervention group will undergo additional Aerobic Training thrice a week for two weeks as well along with postural drainage. Aerobic training will include a 5-step stair-climbing and a 10-step walk during each session. Data will be collected before and at the end of two weeks. Respiratory Rate, Pulse Oximeter, 10-meter Endurance walk test, and Pediatric Cough Questionnaire will be used to collect data pre and post-treatment. Data will be analyzed by use of SPSS Version 2010. Data will be presented in the form of mean and standard deviation.

DETAILED DESCRIPTION:
Chronic suppurative lung disease (csld) is a clinical syndrome in children with respiratory symptoms and signs. Children who have bronchiectasis symptoms but non-diagnostic scans are described as having chronic suppurative lung disease (csld). Postural drainage improves secretion clearance techniques, it is equally as effective as other airway clearance techniques. This study will focus on the implementation of postural drainage and aerobic training in this disease to find their effect on respiratory rate, oxygen saturation, and endurance.

ELIGIBILITY:
Inclusion Criteria:

* Age of 5-13 years
* Medically stable,
* Patients must have 2 episodes of productive cough, each episode lasting for 4 weeks per year.

Exclusion Criteria:

* Non-Chronic Suppurative Lung Disease related chronic disease
* Chronic Suppurative Lung Disease-related conditions posing an increased risk to the patient when exercising.

children with any MSK-disorder or gait abnormalities

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate | 2 weeks
  The respiratory rate is the rate at which breathing occurs; it is set and controlled by the respiratory center of the brain.
Oxygen Saturation | 2 Weeks
  Oxygen saturation is the fraction of oxygen-saturated hemoglobin relative to total hemoglobin in the blood.
10 Meter Walk Test | 2 Weeks
  The individual is instructed to walk a set distance (6 meters, 10 meters, etc). Time is measured while the individual walks the set distance (often the individual is given space to accelerate to his/her preferred walking speed

SECONDARY OUTCOMES:
5-item Pediatric Cough Questionnair | 2 Weeks
  Used to measure frequency of child's cough with aa 6-point Likert-scale. Questionnair have 5 Questions to be answered by parent.

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Altaf, Mphill, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No